CLINICAL TRIAL: NCT03203577
Title: Initiation of Home Mechanical Ventilation at Home in a Selectve Group of Patients With Chronic Hypercapnic Respiratory Failure in the Netherlands
Brief Title: Initiation of Home Mechanical Ventilation at Home in Patients With Chronic Hypercapnic Respiratory Failure
Acronym: Homerun
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Peter Wijkstra, professor, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZonMw 80-83700-98-52003; NTR4683 (Registry Identifier: Dutch trial registry); METc 2014.529 (Other: Medical ethical committee)
Record Dates: First submitted 2017-02-17; First posted 2017-06-29 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Respiratory Therapy; Respiration, Artificial; Positive-Pressure Respiration; Neuromuscular Diseases; Noninvasive Ventilation; Cost-Benefit Analysis; Ambulatory Monitoring
MeSH Terms: conditions — Respiratory Aspiration; Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hospital initiation (Active Comparator): Initiation of mechanical ventilation in hospital initiation of Home Mechanical ventilation takes place in a hospital; this makes this arm the standard care.
  Interventions: Procedure: Initiation of mechanical ventilation
- Home initiation (Experimental): Initiation of mechanical ventilation at home Initiation of mechanical ventilation in a patient's home setting with telemonitoring
  Interventions: Procedure: Initiation of mechanical ventilation

INTERVENTIONS:
Procedure: Initiation of mechanical ventilation — In patient with chronic respiratory insufficient chronic mechanical ventilation will be initiated in the patient his/her setting.
  Other Names: start of home mechanical ventialtion with telemonitoring

SUMMARY:
Objective: To prove that initiation of chronic ventilatory support at home, in patients with chronic hypercapnic respiratory failure due to neuromuscular disease (NMD) or thoracic cage problem is not inferior compared to initiation in a hospital based setting. In addition we believe that the start at home is cheaper compared to an in-hospital start.

Hypothesis: Initiation of chronic ventilatory support at home is effective, safe and cost effective compared to a hospital-based initiation.

Study design: A nationwide non-inferiority multi-center randomized parallel active control study.

Study population: Patients with chronic respiratory insufficiency due to a neuromuscular disease (NMD) or thoracic cage problem who are referred for chronic ventilator support.

Intervention: The start of HMV at home Standard intervention to be compared to: The start of HMV is normally in a clinical setting as recommended in the national guideline.

Outcome measures: Primary: PaCO2. Secondary: Health related quality of life; lung function; nocturnal transcutaneous carbon dioxide assessment and saturation, and costs Sample size calculation/data analysis: This is a non-inferiority trial based on PaCO2 as primary outcome. A difference in favor of the hospital care group of smaller than 0.5 kPa will be labeled as non-inferior. To retain 72 evaluable patients, and allow for drop-outs, we will include 96 patients in total.

Cost-effectiveness analysis: A cost analysis will be conducted alongside the clinical trial. Costs of the initiation of HMV at home and in the hospital will be estimated form a societal perspective over a time horizon of 6 months.

Time schedule: After an initial phase of 6 months recruitment will start and will take 24 months. Thirty-six months after the start of the study the last assessments will be done and analysis and writing of the papers will start. After 42 months the study will end.

ELIGIBILITY:
Inclusion Criteria:

* Indication to initiate non-invasive ventilatory support in patients with a neuromuscular disease or thoracic cage abnormality who suffer from complaints of alveolar hypoventilation (fatigue, headache of dyspnoea) combined with all following elements:
* arterial carbon dioxide > 6.0 kPa daytime or arterial or transcutaneous carbon dioxide > 6.0 kPa at night or orthopnea as a result of diaphragm paralysis
* Age > 18 years
* Existence, of a sufficient network (social or professional) according to the supervising HMV center making initiation of HMV at home possible and safe.

Exclusion Criteria:

* Patients who already have had HMV due to acute respiratory failure
* Necessity for invasive ventilatory support
* Patients admitted to a nursing home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Daytime arterial carbon dioxide | 6 months after initiation of mechanical ventilation
  Daytime arterial carbon dioxide (PaCO2) assessed without oxygen supplementation and ventilatory support while the patient is in sitting position

SECONDARY OUTCOMES:
Quality of life | 6 months after initiation of mechanical ventilation
  Health related quality of life by using the following questionnaires: SF 36, MRF 28, HADS, SRI
Lung function | 6 months after initation of mechanical ventilation
  evaluate lungfunction in time; with measurments of flow/volume in a sitting and horizontal position
Nocturnal transcutaneous carbon dioxide and saturation | 6 months after initiation of mechanical ventilation
  Nocturnal transcutaneous carbon dioxide and saturation in time
costs | 6 months after initiation of mechanical ventilation
  evaluation of the costs during initiation and the follow-up for 6 months. This will be objective by using the EuroQol (EQ-5D) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: P.J. Wijkstra, Prof., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van den Biggelaar RJM, Hazenberg A, Cobben NAM, Gaytant MA, Vermeulen KM, Wijkstra PJ. A Randomized Trial of Initiation of Chronic Noninvasive Mechanical Ventilation at Home vs In-Hospital in Patients With Neuromuscular Disease and Thoracic Cage Disorder: The Dutch Homerun Trial. Chest. 2020 Dec;158(6):2493-2501. doi: 10.1016/j.chest.2020.07.007. Epub 2020 Jul 16. PMID 32682770